CLINICAL TRIAL: NCT04359095
Title: Effectiveness and Safety of Medical Treatment for SARS-CoV-2 (COVID-19) in Colombia: A Pragmatic Randomized Controlled Trial
Brief Title: Effectiveness and Safety of Medical Treatment for SARS-CoV-2 (COVID-19) in Colombia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Pontificia Universidad Javeriana (Other); Clínica Colsanitas-Clínica Universitaria Colombia (Unknown); Hospital Universitario San Ignacio (Other); Hospital Universitario Nacional de Colombia (HUN) (Unknown); Fundación Cardioinfantil Instituto de Cardiología (Other); Clínica Infantil Santa María del Lago (Unknown)
Responsible Party: Principal Investigator, Hernando Gaitán, MD, Professor at the Obstetrics and Gynecology Department and Clinical Research Institute. Director of Research and Extension in the Bogota Campus at The Universidad Nacional de Colombia, Co- Ed. Sexually Transmitted Infections Cochrane Review Group, Universidad Nacional de Colombia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76968
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: COVID-19; COVID-19 drug treatment
MeSH Terms: conditions — COVID-19 | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Colchicine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- I1 Emtricitabine + Tenofovir (Active Comparator): Intervention 1: Emtricitabine (200 mg) + tenofovir (300 mg): 500 mg once a day for 10 days
  Interventions: Drug: Emtricitabine/tenofovir
- I2 Colchicine + rosuvatatine (Active Comparator): Intervention 2: Colchicine: 0.5 mg every 12 hours for 14 days + Rosuvatatin: 40 mg / day for 14 days
  Interventions: Drug: Emtricitabine/tenofovir; Drug: Colchicine Pill
- I3 Emtricitabine/ tenofobir + colchicine+ rosuvastatin (Active Comparator): Intervention 3: Emtricitabine (200 mg) + tenofovir (300 mg): 500 mg once a day for 10 days + Colchicine: 0.5 mg every 12 hours for 14 days + Rosuvatatin: 40 mg / day for 14 days
  Interventions: Drug: Emtricitabine/tenofovir; Drug: Rosuvastatin
- I4 Standard Treatment (Other): Intervention 4: Standard treatment. It is defined as treatment aimed to control symptoms including fever and pain, multiple organ failure related to the acute infection including respiratory support (oxygen, positive end-expiration pressure with external devices or invasive ventilatory support), cardiovascular, renal, haematological or coagulation, or co-infection with bacterial or mycotic organisms, standard care to prevent pressure ulcers or other care required by the patient, might include Dexamethasone. No viral therapies are included.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Drug: Emtricitabine/tenofovir — Generic drug distributed by the Colombian Health System for Human Immunodeficiency Virus (HIV) positive patients It is classified as an anti infectious drug and its current indications include HIV infections.
  Other Names: Truvada ®
  Arms: I1 Emtricitabine + Tenofovir; I2 Colchicine + rosuvatatine; I3 Emtricitabine/ tenofobir + colchicine+ rosuvastatin
Drug: Colchicine Pill — Generic drug distributed by the Colombian Health System as an insurance treatment for Gout. It has been suggested that colchicine would be useful in SARS Covid 19 becouse its antiinflammatory effects through reduction of cytokine levels as well as the activation of macrophages, neutrophils, and the inflammasome
  Arms: I2 Colchicine + rosuvatatine
Drug: Rosuvastatin — Generic drug distribute by the Colombian Health System. It is used in people with High levels of cholesterol. An action against the main protease (Mpro) of COVID 19 virus has been described, There is evidence suggesting that statins could exert anti Covid 19 action and the infectivity of enveloped viruses
  Other Names: Crestor ® Rosuvas ®
  Arms: I3 Emtricitabine/ tenofobir + colchicine+ rosuvastatin
Other: Standard treatment — Standard treatment n, multiple organ failure related to the acute infection including respiratory support (oxygen, positive end-expiration pressure with external devices or invasive ventilatory support), cardiovascular, renal, haematological or coagulation, or co-infection with bacterial or mycotic organisms, standard care to prevent pressure ulcers or other care required by the patient. No viral therapies are included.
  Arms: I4 Standard Treatment

SUMMARY:
Introduction: The COVID-19 pandemic is characterized by significant morbidity and mortality. Treatments have been administered to patients with COVID-19 in order to control viral infection, among them: Hydroxychloroquine (HCQ), Lopinavir/Ritonavir (Lop/r), Remdesivir, Favipavir, Emtricitabine/ Tenofovir acting over bacterial co-infection Azithromycin (Azithro), or modifying the inflammatory response of the host (Tocilizumab, colchicine, dexamethasone, and by other mechanisms (rosuvastatin). Except for dexamethasone clinical trials offer conflicting evidence regarding the effectiveness and safety of therapies.

Objective: Evaluate the effectiveness and safety of pharmacological therapies used to treat adult patients with COVID-19.

Methods: Pragmatic randomized controlled trial. Study population: Adults aged 18 years or over with a positive real-time polymerase chain reaction (RT-PCR) or with high suspicion of Severe Acute Respiratory Syndrome CoV-2 (SARS CoV-2) and diagnosis of mild, severe or critical pneumonia, requiring hospital management at six hospitals in Colombia. Exclusion criteria: Pregnancy, known allergy to treatment, cirrhosis or hepatic abnormality (transaminases greater than 5 reference values), glomerular filtration rate lesser than 30 ml/min/1.73m^2, history of lung fibrosis, advanced or metastatic cancer. A sample size was calculated from a sensitivity analysis with three scenarios:

scenario 1 a total of 1,163 patients, that is, 291 per treatment arm with alpha of Alpha = 0.05; power 0.8; Prop1 = 0.2 and Prop2 = 0.1 (expected difference of 10%) and 10% of possible losses,scenario 2. With the previous parameters and with a Prop1 = 0.15 and Prop2 = 0.05 for a total of 814 patients (204 per arm of treatment). scenario 3. With Alpha = 0.1, Prop1 = 0.15 and Prop2 = 0.05, the other previous parameters, for a total of 686 patients (172 per treatment). in scenario 1 the study will be carried out in two phases. The first phase will be conducted with 400 participants and aims to identify treatments with higher or minimum potential, discontinue treatments with higher toxicity, and have the opportunity of introducing new treatments with potential efficacy. The second phase will be conducted with 1,163 participants to evaluate the effectiveness of the selected treatments.

Four interventions have been defined: I1 Emtricitabine/ teneofovir , I2 Colchicine plus rosuvastatin, I3 Emtricitabine/ teneofovir plus Colchicine plus rosuvastatin and I4 standard treatment. Within each institution, participants will be randomly assigned to one of the treatment arms assigned to that institution. Concealment will be kept through software that maintain the assignment concealed until the random assignment is done . Treatment administration will be open. Variables: Sociodemographic and clinical at recruitment; (comorbidities, need for therapeutic support , grade of invasion at admission). Primary outcomes. Effectiveness: Mortality. Safety: Serious adverse events (AE) assessed by the NCI Community Oncology Research Program (NCORP) Guidance for Collection of Adverse Events Related to COVID-19 Infection. Secondary outcomes: Intensive care unit (ICU) admission, requirement of respiratory support, time to death, number of participants cured, any adverse event related to treatment.

Analysis: Descriptive for the presentation of summary measures of the basal conditions by type of variable. Bivariate. Description of the basal conditions (with organic failure at admission, without failure at admission), by type of treatment, by participating institution. Description of crude effectiveness and safety by means of the difference of accumulated incidences, each one with 95% confidence intervals (95% CI) Intention to treat analyisis will be done. Adjusted analysis: The ratio and difference of cumulative incidences of mortality at 7 and 28 days and severe adverse events between treatments will be estimated, adjusting for confounding variables using logistic regression models with mixed effects considering each institution as a level or from equations. generalized estimation (GEE). On the other hand, as part of the pragmatic approach, the surface under cumulative ranking curve (SUCRA) will be calculated based on Bayesian theory to define which drug has the highest probability of being the most useful in the management of infection.

Ethical considerations: The study has a risk beyond minimum according to the Resolution 8430/1993 of the Colombian Ministry of Health. Informed consent will be explained and signed if the patient is in condition to do so. This protocol will undergo evaluation by the ethics committee at each of the participating institutions and at the National University of Colombia. The protocol follows the Helsinki Declaration and institutional protocols for clinical investigation.

DETAILED DESCRIPTION:
Initially, the use of the drugs chloroquine, hydroxychloroquine and lopinavir / ritonavir had been proposed in this study, based on laboratory results of their in vitro antiviral potency for the CoV-2 virus, but with limited clinical evidence. However, later there were problems with the safety of the use of azithromycin in patients with SARS Covid 19. The coordinating committee of this study decided by consensus to suspend the use of hydroxychloroquine in the clinical trial in question by means of minutes of June 9, 2020 given that the interim analysis of the Recovery study showed (on June 5) that "there are no differences between hydroxychloroquine and standard treatment (28-day mortality between HCQ hydroxychloroquine and standard treatment (28-day mortality outcome (25.7% hydroxychloroquine vs. 23.5% usual care; Hazard ratio (HR: 1.11 [95% CI 0.98-1.26]). "(21) On the other hand, on June 29, the same Recovery study published the results of the interim analysis on the use of lopinavir ritonavir in patients with SARS Covid 19. In a statement it reports that "there were no significant differences in the 28-day mortality outcome (22.1% of lopinavir-ritonavir versus 21.3 % of usual care; (relative risk RR 1.04 95% CI 0.91-1.18]; no beneficial effects were found on the risk of progression to mechanical ventilation or the length of hospital stay "(22)

Given these results, it is relevant to know the clinical effectiveness and adverse effects of the drugs: emtricitabine / tenofovir, colchicine / rosuvastatin, compared with the usual management, as alternatives for the management of COVID-19 infection in real patient scenarios for support decision making in clinical practice.

Interim analysis and sample size

A sample size was calculated from a sensitivity analysis with three scenarios:

scenario 1 a total of 1,163 patients, that is, 291 per treatment arm with alpha of Alpha = 0.05; power 0.8; Prop1 = 0.2 and Prop2 = 0.1 (expected difference of 10%) and 10% of possible losses, scenario 2. With the previous parameters and with a Prop1 = 0.15 and Prop2 = 0.05 for a total of 814 patients (204 per arm of treatment) scenario 3. With Alpha = 0.1, Prop1 = 0.15 and Prop2 = 0.05, the other previous parameters, for a total of 686 patients (172 per treatment).

A sample size was calculated from a sensitivity analysis with three scenarios:

scenario 1 a total of 1,163 patients, that is, 291 per treatment arm with alpha of Alpha = 0.05; power 0.8; Prop1 = 0.2 and Prop2 = 0.1 (expected difference of 10%) and 10% of possible losses, scenario 2. With the previous parameters and with a Prop1 = 0.15 and Prop2 = 0.05 for a total of 814 patients (204 per arm of treatment) scenario 3. With Alpha = 0.1, Prop1 = 0.15 and Prop2 = 0.05, the other previous parameters, for a total of 686 patients (172 per treatment)

Under this new approach we will make an evaluation of the minimum effectiveness in scenarios 1 and 2 :

Stage 1 When completing the sample size of this stage (400 participants), a interim analysis will be carried out that allows testing whether there is an expected difference of 15 percent (25 percent - 10 percent), with a power of 84 percent. As in the previous analysis, if significant differences are found, the treatment with less effectiveness (highest mortality) is replaced. The correction of the type I error will be made using the O'Brien-Fleming method.

Stage 2. Estimation of effectiveness:

When we have a sample size of 290 participants in each intervention, allowing the evaluation of an expected difference of 10 (20percent - 10 percent) with a power of 81 percent and a significance level of 0.05. A loss percentage of 10 will be considered.

Rules for selecting a drug to be included in the RCT in stage 1

Criteria for inclusion of a new drug, in its order:

1. Evidence that the drug is safe in humans
2. The drug must have a record from the National Institute for Food and Drug Surveillance (Invima)
3. Drug's availability in the country
4. The drug must show at least 15 percent superiority to standard management in other randomized clinical trials that have been conducted in patients with SARS CoV-2 / COVID-19
5. Biological plausibility and studies that support the choice: in vitro case series studies, use in similar situations
6. Ongoing studies that are evaluating the drug's effectiveness and safety
7. The drug must meet the objective of the study

In the scenario 2 and 3 we will no do an interim analysis

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for institutions:

* Centralized pharmacy department which allows safe storage of drugs
* Centralized pharmacy department that follows good clinical practice protocols for investigation

and either

* ICU capacity of at least 10 beds with available ventilatory support (volume) or
* Intermediate care unit with at least 10 beds with partial ventilatory support

Inclusion criteria for participants:

- Age 18 years or over

- Positive RT-PCR for COVID-19 or high suspicion of SARS covid 19

- Requirement of in-hospital treatment, classified in any of the following categories:

1. Mild pneumonia, defined as:

   - Confirmed pneumonia with chest X-Rays

   and at least 2 of the following risk factors or complications:
   * Age 60 years or over
   * History of cardiovascular disease
   * History of diabetes mellitus (DM)
   * History of chronic obstructive pulmonary disease (COPD)
   * History of hypertension (HT)
   * Cancer

   or
2. Moderate pneumonia, defined as :

   - Confirmed pneumonia with chest X-Rays

   and either

   - Criteria for in-hospital management according to the simplified confusion- respiratory rate- blood pressure- age scale (CRB-65 scale) score greater than 1 or Oxygen saturation lower than 90 percent without supplementary oxygen.

   or
3. Severe pneumonia, sepsis or septic shock, defined as:

   * Confirmed pneumonia with chest X-Rays and either
   * Criteria for in-hospital management according to the simplified CRB-65 scale (score greater than 1) or
   * Oxygen saturation lower than 90 percent without supplementary oxygen

and any of the following:

* Respiratory rate greater than 30 per minute
* Need for mechanical ventilation (invasive or non-invasive)
* Sepsis defined as organic dysfunction which can be identified by a Sequential Organ Failure Assessment score (SOFA score) of at least 2 points
* Quick sequential organ failure assessment score (qSOFA) score with 2 of the following criteria:
* Glasgow of 13 or lower, systolic blood pressure of 100 mmHg or lower and respiratory rate equal to or higher than 22 per minute
* Arterial hypotension which persists after hydric resuscitation and requires vasopressors to maintain a mean arterial pressure greater than 65 mmHg and lactate lesser than 2 mmol/L (18 mg/dL) without hypovolemia (referred as septic shock)
* Multiple organ failure
* Acute Respiratory Distress Syndrome (radiological findings compatible with bilateral infiltrates and oxygenation deficit classified as: mild (PaO2/FiO2 between 200 and 300), moderate (PaO2/FiO2 between 100 and 200) or severe (PaO2/FiO2 lower than 100)).

Exclusion Criteria for participants:

* Pregnancy
* Known allergies to the drugs under study
* Hepatic cirrhosis (Child B or C) or hepatic abnormality manifested as transaminase levels 5 times above reference values
* Glomerular filtration rate lesser than 30 ml/min/1.73^m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Advanced or metastatic cancer
* Fatigue, Resistance, Ambulation, Illnesses, and Loss of weight questionnaire (FRAIL) score of fragility greater than 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality | Post-intervention at day 28
  Cumulative incidence
Number of Participants with Treatment Related Severe Adverse Events as Assessed by the NCORP Guidance for Collection of Adverse Events Related to COVID-19 Infection | Post-intervention at day 28
  Number of participants that develop severe adverse events related to the treatment

SECONDARY OUTCOMES:
Mortality | Post-intervention at day 7
  Cumulative incidence
Number of Participants with Treatment Related Severe Adverse Events as Assessed by the NCORP Guidance for Collection of Adverse Events Related to COVID-19 Infection | Post-intervention at day 7
  Number of participants that develop severe adverse events related to the treatment
Time to death | Assessed up to 28 days postintervention
  Time from the date of assignment until the date of death from any cause
Number of Participants that are transferred to the Intensive Care Unit (ICU) | Post-intervention at day 28
  Number of Participants that require management in the ICU
Number of Participants that need Mechanical Ventilation Support with endotracheal intubation. | Up to 28 days after hospital admission
  Participants requiring invasive mechanical ventilation
Number of participants Cured assessed by Nasopharyngeal swab, oropharyngeal swab, and blood aspiration for COVID19 (RT-PCR) without clinical symptoms and normal chest X ray | Up to 28 days after hospital admission
  Number of participants cured assessed RT-PCR for SARS CoV-2, without clinical symptoms and no radiological signs assessed by chest X ray
Number of Participants with Any Adverse Event Related to Treatment Assessed by the NCORP Guidance for Collection of Adverse Events Related to COVID-19 Infection | Up to 28 days after hospital admission
  Any adverse event

OTHER OUTCOMES:
Severe Adverse events | Up to 28 days after hospital admission
  Interim assessment of safety, which will be conducted after 400 number of participants with severe adverse events divided by the total number of participants treated). It aims to aid the decision of excluding an active treatment arm should that arm have more than 3 serious adverse events in the first 30 participants or a serious adverse events incidence of 10 percent or higher.
Mortality | Up to 28 days after hospital admission
  Interim assessment of minimum effectiveness, which will be conducted after 480 participants are recruited. It will be evaluated through relative frequency measurements (mortality proportion at 28 days of treatment). It aims to aid the decision of excluding an active treatment arm should that treatment arm have an efficacy lower than 0.2, calculated through futility analysis that assumes an expected difference of 10 percent at the end of the first phase of the study. For all the tests carried out in the interim analysis, the correction of the type I error will be made using the O'Brien-Fleming method.

CONTACTS AND LOCATIONS:
Overall Officials: Hernando Gaitán, MD, Principal Investigator — Universidad Nacional de Colombia
Locations (6):
- Colombia (6):
  - Clinica santa Maria del lago, Bogotá, DC
  - Clínica Reina Sofía, Bogotá
  - Fundacion Cardio Infantil, Bogotá
  - Hospital Universitario San Ignacio, Bogotá
  - Clinica Universitaria Colombia, Bogotá
  - Hospital Universitario Nacional de Colombia, Bogotá

IPD SHARING:
Plan to Share IPD: Yes
Communicating trial results and data to be able to combine data from multiple studies (live SR)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon we have checked the quality of data of recruited participants
Access Criteria: Approved by the monitor committee of the study

REFERENCES:
- [Result] Hatem A, Mohamed S, Abu Elhassan UE, Ismael EAM, Rizk MS, El-Kholy A, El-Harras M. Clinical characteristics and outcomes of patients with severe acute respiratory infections (SARI): results from the Egyptian surveillance study 2010-2014. Multidiscip Respir Med. 2019 Apr 1;14:11. doi: 10.1186/s40248-019-0174-7. eCollection 2019. PMID 30976418
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Munster VJ, Koopmans M, van Doremalen N, van Riel D, de Wit E. A Novel Coronavirus Emerging in China - Key Questions for Impact Assessment. N Engl J Med. 2020 Feb 20;382(8):692-694. doi: 10.1056/NEJMp2000929. Epub 2020 Jan 24. No abstract available. PMID 31978293
- [Result] Zu ZY, Jiang MD, Xu PP, Chen W, Ni QQ, Lu GM, Zhang LJ. Coronavirus Disease 2019 (COVID-19): A Perspective from China. Radiology. 2020 Aug;296(2):E15-E25. doi: 10.1148/radiol.2020200490. Epub 2020 Feb 21. PMID 32083985
- [Result] Asociación Colombiana de Infectología. Consenso Colombiano de atención, diagnóstico y manejo de la Infección por SARS COV-2 / COVID 19 en establecimientos de atención de la salud. 2020.
- [Result] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Result] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Result] Mo Y, Fisher D. A review of treatment modalities for Middle East Respiratory Syndrome. J Antimicrob Chemother. 2016 Dec;71(12):3340-3350. doi: 10.1093/jac/dkw338. Epub 2016 Sep 1. PMID 27585965
- [Result] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Result] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Result] Romanelli F, Smith KM, Hoven AD. Chloroquine and hydroxychloroquine as inhibitors of human immunodeficiency virus (HIV-1) activity. Curr Pharm Des. 2004;10(21):2643-8. doi: 10.2174/1381612043383791. PMID 15320751
- [Result] Yan Y, Zou Z, Sun Y, Li X, Xu KF, Wei Y, Jin N, Jiang C. Anti-malaria drug chloroquine is highly effective in treating avian influenza A H5N1 virus infection in an animal model. Cell Res. 2013 Feb;23(2):300-2. doi: 10.1038/cr.2012.165. Epub 2012 Dec 4. No abstract available. PMID 23208422
- [Result] Khan M, Santhosh SR, Tiwari M, Lakshmana Rao PV, Parida M. Assessment of in vitro prophylactic and therapeutic efficacy of chloroquine against Chikungunya virus in vero cells. J Med Virol. 2010 May;82(5):817-24. doi: 10.1002/jmv.21663. PMID 20336760
- [Result] Farias KJ, Machado PR, de Almeida Junior RF, de Aquino AA, da Fonseca BA. Chloroquine interferes with dengue-2 virus replication in U937 cells. Microbiol Immunol. 2014 Jun;58(6):318-26. doi: 10.1111/1348-0421.12154. PMID 24773578
- [Result] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Result] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Result] Ruuskanen O, Lahti E, Jennings LC, Murdoch DR. Viral pneumonia. Lancet. 2011 Apr 9;377(9773):1264-75. doi: 10.1016/S0140-6736(10)61459-6. Epub 2011 Mar 22. PMID 21435708
- [Result] de Wit E, van Doremalen N, Falzarano D, Munster VJ. SARS and MERS: recent insights into emerging coronaviruses. Nat Rev Microbiol. 2016 Aug;14(8):523-34. doi: 10.1038/nrmicro.2016.81. Epub 2016 Jun 27. PMID 27344959
- [Result] Short KR, Kedzierska K, van de Sandt CE. Back to the Future: Lessons Learned From the 1918 Influenza Pandemic. Front Cell Infect Microbiol. 2018 Oct 8;8:343. doi: 10.3389/fcimb.2018.00343. eCollection 2018. PMID 30349811
- [Result] Lipatov AS, Govorkova EA, Webby RJ, Ozaki H, Peiris M, Guan Y, Poon L, Webster RG. Influenza: emergence and control. J Virol. 2004 Sep;78(17):8951-9. doi: 10.1128/JVI.78.17.8951-8959.2004. No abstract available. PMID 15308692
- [Result] Remolina YA, Ulloa MM, Vargas H, Diaz L, Gomez SL, Saavedra A, Sanchez E, Cortes JA. Viral Infection in Adults with Severe Acute Respiratory Infection in Colombia. PLoS One. 2015 Nov 17;10(11):e0143152. doi: 10.1371/journal.pone.0143152. eCollection 2015. PMID 26576054
- [Result] Lachin JM. A review of methods for futility stopping based on conditional power. Stat Med. 2005 Sep 30;24(18):2747-64. doi: 10.1002/sim.2151. PMID 16134130
- [Derived] Gaitan-Duarte HG, Alvarez-Moreno C, Rincon-Rodriguez CJ, Yomayusa-Gonzalez N, Cortes JA, Villar JC, Bravo-Ojeda JS, Garcia-Pena A, Adarme-Jaimes W, Rodriguez-Romero VA, Villate-Soto SL, Buitrago G, Chacon-Sarmiento J, Macias-Quintero M, Vaca CP, Gomez-Restrepo C, Rodriguez-Malagon N. Effectiveness of rosuvastatin plus colchicine, emtricitabine/tenofovir and combinations thereof in hospitalized patients with COVID-19: a pragmatic, open-label randomized trial. EClinicalMedicine. 2022 Jan;43:101242. doi: 10.1016/j.eclinm.2021.101242. Epub 2021 Dec 20. PMID 34957385